CLINICAL TRIAL: NCT00652340
Title: APRiCOT-L (Apricoxib in Combination Oncology Treatment - Lung) A Randomized, Double-Blind, Placebo-Controlled Multicenter Phase 2 Study of the Efficacy and Safety of Apricoxib in Combination With Erlotinib in Non-Small Cell Lung Cancer Patients
Brief Title: APRiCOT-L: Study to Evaluate Efficacy and Safety of Apricoxib With Erlotinib in Patients With Non-small Cell Lung Cancer
Acronym: TP2001-201
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tragara Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TP2001-201; APRiCOT-L
Record Dates: First submitted 2008-03-31; First posted 2008-04-03 (Estimated); Results first posted 2012-04-09 (Estimated); Last update posted 2012-04-09 (Estimated); Status verified 2012-03

CONDITIONS: Recurrent Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — apricoxib; Erlotinib Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental)
  Interventions: Drug: apricoxib/erlotinib
- B (Placebo Comparator)
  Interventions: Drug: erlotinib/placebo

INTERVENTIONS:
Drug: apricoxib/erlotinib — apricoxib: 100 mg tablets, 400mg/day
  erlotinib: per package insert
  Arms: A
Drug: erlotinib/placebo — erlotinib: per package insert
  placebo: 100 mg tablets, 400 mg/day
  Arms: B

SUMMARY:
This study will compare the anti-tumor efficacy of apricoxib and erlotinib with placebo and erlotinib as measured by time to disease progression to test the hypothesis that down regulation of COX-2 and EGFR pathways in patients with up-regulated COX-2 expression in tumor will have a clinical benefit compared with erlotinib alone.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically determined Stage IV NSCLC including Stage IIIb (pleural effusion)
* Failed at least one prior platinum-based chemotherapy for Stage IIIb or Stage IV NSCLC. Patients receiving platinum-based chemotherapy only given in an adjuvant setting are not eligible.
* Measurable disease by RECIST
* Greater than or equal to 18 years of age
* ECOG PS of 0 or 1

Exclusion Criteria:

* Radiation therapy within 2 weeks; chemotherapy within 3 weeks; non-cytotoxic investigational agents within 4 weeks of initiating study treatment
* Evidence of NYHA class III or greater cardiac disease
* History of MI, stroke, ventricular arrhythmia, or symptomatic conduction abnormality within 12 months
* Known HIV infection or AIDS
* Symptomatic CNS metastases
* Pregnant or nursing women
* Hypersensitivity or intolerance to erlotinib, sulfonamides, aspirin, or other NSAIDs.
* History of upper GI bleeding, ulceration, or perforation
* Prior history of COX-2 inhibitor therapy for the treatment of metastatic NSCLC
* Previous anti-EGFR kinase therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2008-04; Primary Completion 2010-06 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tracy Parrott, Study Director — Tragara Pharmaceuticals, Inc.
Locations (47):
- United States (47):
  - Tucson, Arizona
  - Bakersfield, California
  - Los Angeles, California
  - Rancho Mirage, California
  - San Diego, California
  - San Dimas, California
  - Stockton, California
  - Norwich, Connecticut
  - Lake North, Florida
  - Lakeland, Florida
  - Miami, Florida
  - Savannah, Georgia
  - Chicago, Illinois
  - Kokomo, Indiana
  - New Albany, Indiana
  - Waterloo, Iowa
  - Louisville, Kentucky
  - New Orleans, Louisiana
  - Ann Arbor, Michigan
  - Jackson, Michigan
  - Lansing, Michigan
  - Livonia, Michigan
  - Saginaw, Michigan
  - Saint Joseph, Michigan
  - Robbinsdale, Minnesota
  - St Louis, Missouri
  - Neptune City, New Jersey
  - Elmhurst, New York
  - Stony Brook, New York
  - Gastonia, North Carolina
  - Wilmington, North Carolina
  - Akron, Ohio
  - Canton, Ohio
  - Columbus, Ohio
  - Jefferson, Ohio
  - Sylvania, Ohio
  - Corvallis, Oregon
  - Portland, Oregon
  - Upland, Pennsylvania
  - Charleston, South Carolina
  - Arlington, Texas
  - Galveston, Texas
  - Newport News, Virginia
  - Richmond, Virginia
  - Tacoma, Washington
  - Huntington, West Virginia
  - Morgantown, West Virginia

REFERENCES:
- [Derived] Gitlitz BJ, Bernstein E, Santos ES, Otterson GA, Milne G, Syto M, Burrows F, Zaknoen S. A randomized, placebo-controlled, multicenter, biomarker-selected, phase 2 study of apricoxib in combination with erlotinib in patients with advanced non-small-cell lung cancer. J Thorac Oncol. 2014 Apr;9(4):577-82. doi: 10.1097/JTO.0000000000000082. PMID 24736085

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study opened to accural in April 2008. Enrollment closed in May 2010. One hundred seventy six patients were enrolled with 120 patients randomized. Patients were recruited from clinical oncology practices.
Pre-assignment Details: Enrolled patients underwent a 5-day open label treatment with apricoxib to determine the maximum suppression of PGEM from a baseline measurment. PGEM was used as a biomarker of COX-2 activity in the tumor. Patients with at least a 50% decrease on day 5 from their baseline measurment were eligible to be randomized.
Groups:
- Apricoxib/Erlotinib: Patients randomized to receive apricoxib and erlotinib.
- Placebo/Erlotinib: Patients randomized to receive placebo and erlotinib.
Period: Overall Study
Arm/Group | Apricoxib/Erlotinib | Placebo/Erlotinib
Started | 78 | 42
Completed | 74 (4 patients remained on study at database lock.) | 39 (3 patients remained on study at database lock.)
Not Completed | 4 | 3
Not completed — Had not progressed. | 4 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Apricoxib/Erlotinib | Placebo/Erlotinib | Total
Number analyzed (Participants) | 78 | 42 | 120
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 46 | 23 | 69
  >=65 years | 32 | 19 | 51
Age Continuous [Mean (Standard Deviation); unit: years] | 62.1 (10.78) | 64.6 (11.16) | 62.9 (10.94)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 17 | 53
  Male | 42 | 25 | 67
Region of Enrollment [Number; unit: participants]
  United States | 78 | 42 | 120

OUTCOME MEASURES:

1. Primary Outcome: Time to Disease Progression (TDP)
Time Frame: Baseline and every other cycle.
Population: A 1-sided log rank test was used to achieve 80% power at an α=0.20 significance level to detect a difference of 0.13 between the proportions of patients who are progression free in AP/E (0.34) and P/E (0.21) after 5 months; an overall sample size of 115 patients (77 in AP/E and 38 in P/E) will be randomized in a 2:1 ratio in this study.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Apricoxib/Erlotinib | Placebo/Erlotinib
Number analyzed (Participants) | 78 | 42
months | 1.80 [1.40 to 2.80] | 2.10 [1.40 to 4.00]

2. Secondary Outcome: Overall Survival
Time Frame: Randomization and every cycle
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Apricoxib/Erlotinib | Placebo/Erlotinib
Number analyzed (Participants) | 78 | 42
months | 5.90 [4.10 to 8.50] | 5.60 [3.80 to 9.10]

ADVERSE EVENTS:
Time Frame: First dose of study drug to 30 days after last dose of study drug.
Description: Only drug related serious adverse events are listed.
Arm/Group | Apricoxib/Erlotinib | Placebo/Erlotinib
Serious Adverse Events (participants affected / at risk) | 13/78 | 4/42
Other Adverse Events (participants affected / at risk) | 77/78 | 42/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Apricoxib/Erlotinib (N=78) | Placebo/Erlotinib (N=42)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Left ventricular dysfunction (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Gastric ulcer perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1)
Intestinal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Peritonitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 1 (1) | 0 (0)
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Apricoxib/Erlotinib (N=78) | Placebo/Erlotinib (N=42)
Rash (Skin and subcutaneous tissue disorders) | 42 (42) | 23 (23)
Diarrhea (Gastrointestinal disorders) | 41 (41) | 25 (25)
fatigue (General disorders) | 33 (33) | 12 (12)
Nausea (Gastrointestinal disorders) | 27 (27) | 12 (12)
Dry skin (Skin and subcutaneous tissue disorders) | 20 (20) | 11 (11)
Cough (Respiratory, thoracic and mediastinal disorders) | 18 (18) | 5 (5)
Anorexia (General disorders) | 17 (17) | 15 (15)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 16 (16) | 11 (11)
Vomiting (Gastrointestinal disorders) | 16 (16) | 4 (4)
Mucosal inflammation (Gastrointestinal disorders) | 15 (15) | 4 (4)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 13 (13) | 11 (11)
Constipation (Gastrointestinal disorders) | 12 (12) | 5 (5)
Insomnia (Psychiatric disorders) | 11 (11) | 7 (7)
Dizziness (Nervous system disorders) | 10 (10) | 4 (4)
Dyspepsia (Gastrointestinal disorders) | 10 (10) | 6 (6)
Pruritis (Skin and subcutaneous tissue disorders) | 10 (10) | 9 (9)
Anemia (Blood and lymphatic system disorders) | 9 (9) | 2 (2)
Blood creatinine increased (Investigations) | 9 (9) | 0 (0)
Weight decreased (General disorders) | 9 (9) | 6 (6)
Edema peripheral (Musculoskeletal and connective tissue disorders) | 8 (8) | 6 (6)
Anxiety (Psychiatric disorders) | 7 (7) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 7 (7) | 5 (5)
Dehydration (General disorders) | 7 (7) | 3 (3)
Epistaxis (Skin and subcutaneous tissue disorders) | 7 (7) | 1 (1)
Pneumonia (Infections and infestations) | 7 (7) | 4 (4)
Alopecia (Skin and subcutaneous tissue disorders) | 6 (6) | 4 (4)
Depression (Psychiatric disorders) | 6 (6) | 2 (2)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 5 (5) | 5 (5)
Dysgeusia (Gastrointestinal disorders) | 5 (5) | 3 (3)
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 2 (2)
Hypertension (Cardiac disorders) | 5 (5) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days